CLINICAL TRIAL: NCT03048773
Title: Extracorporeal Shockwave Therapy for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TYGH105013
Record Dates: First submitted 2017-01-24; First posted 2017-02-09 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Shockwave Therapy; Knee Osteoarthritis
Keywords: shockwave therapy; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shockwave therapy (Experimental): 1. 0.24mJ/mm2，1600 shots over 8 assigned sites of single knee with jelly between applicator pad (20) and handpiece
  2. Physical therapy with TENS + MF + stretching + strengthening exercise, 3 times per week for 3 weeks
  Interventions: Device: shockwave therapy; Other: PT
- placebo (Placebo Comparator): 1. 0.24mJ/mm2，1600 shots over 8 assigned sites of single knee without jelly between applicator pad (20) and handpiece
  2. Physical therapy with TENS + MF + stretching + strengthening exercise, 3 times per week for 3 weeks
  Interventions: Other: PT; Other: placebo

INTERVENTIONS:
Device: shockwave therapy — Intervention with shockwave therapy
  Arms: shockwave therapy
Other: PT — Physical therapy 3 times per week for 3 weeks
Other: placebo — sham shockwave therapy
  Arms: placebo

SUMMARY:
Knee osteoarthritis is a common disease that causes joint pain, stiffness, and movement limitation. Nearly 50% in those 75 years and above are affected. In Taiwan, the reported prevalence was more than 6000 per year. The cause of pain is joint instability and structure changed, including hyaline articular cartilage lost, bony remodeling, capsular stretching and periartcular muscle weakness. Current guidelines for treatment of symptomatic knee osteoarthritis include exercise, anti-inflammatory drugs, transcutaneous electrical stimulation(TENS) and magnetic fields(MF) which reduce pain and improve the patient's quality of life.

However, conservative therapies and oral supplements have been evaluated but are without clear efficacy. Prolotherapy is an injection therapy for chronic musculoskeletal pain. One of the hypotheses is stimulating local healing and current study demonstrated clinical benefit for pain and improvement of function. The effects of multi-point injections were more pronounced in several studies than single-point injection.

Extracorporeal shock wave is common treatment for kidney stones, has been widely used in soft tissue diseases, such as calcified tendon lesions and plantar fasciitis. The theory of extracorporeal shock wave is energy of high-frequency vibration caused destruction of stones and other hard material and by increasing the rate of vascular regeneration in the injured area and increasing the rate of autologous tissue repair, possible biological processes include increased mesenchymal stem cell proliferation and differentiation, slowing the inflammatory response and antimicrobial efficacy. Current studies have shown equivalent clinical outcomes on calcific rotator cuff tendinopathy among extracorporeal shock wave therapy, sono-guided acupuncture and arthroscopic surgery and the extracorporeal shock wave has the advantage of non-invasive treatment.

Taking the advantages of non-invasive treatment of extracorporeal shockwave. We want to design a randomized control trial by multi-point shockwave therapy and physical therapy compared with placebo shockwave therapy and physical therapy. Two randomized controlled trial (RCT) reported improvement in outcomes in response to shockwave therapy but were not methodologically rigorous. The investigators therefore conducted a two-arm RCT to assess the hypothesis that adults with symptomatic knee pain receiving shockwave therapy will report greater improvement in knee-related quality-of-life than sham shockwave therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient at Taoyuan general hospital rehabilitation outpatient department during 2017/01/01 ~ 2018/12/31
2. Diagnosis with knee osteoarthritis (ACR criteria or Kellgren and Lawrence grading II to IV)
3. Suitable for shockwave therapy and physical therapy with (TENS + MF + stretching + strengthening exercise)
4. Visual analog scale(VAS) ≧ 4

Exclusion Criteria:

1. Not suitable for shockwave therapy, including acute infection, osteomyelitis, coagulopathy, use of anticoagulants, pregnant women, patients with a pacemaker or implantable cardiac defibrillator
2. Patients who can't understand Chinese, including aphasia or dementia
3. Patient who can't receive 4 weeks of therapy
4. Patient who can't walk due to peripheral neuropathy or central nerve system diseases
5. Total knee arthroplasty
6. Shockwave therapy of knee for the prior 3 months
7. Skin defect or soft tissue infection over symptomatic knee
8. Other cause of knee pain which can't treat with physical therapy, including: rheumatoid arthritis, infection, fracture, ligament disruption

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
WOMAC score by Chinese version NRS 3.1 | Change from baseline to week 3 and week 4
six minute walk test | Change from baseline to week 3 and week 4
  The distance covered in meters of six minute walk test

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Change from baseline to week 3 and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Huan-Jui Yeh, Principal Investigator — Taoyuan General Hospital
Locations (1):
- Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho KD, Yang CL, Lo HY, Yeh HJ. Extracorporeal Shockwave Therapy With a Modified Technique on Tendon and Ligament for Knee Osteoarthritis: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Jan 1;101(1):11-17. doi: 10.1097/PHM.0000000000001730. PMID 34915541